CLINICAL TRIAL: NCT01153659
Title: A Randomized, Open-Label, Three-Way Crossover Study to Evaluate the Effect on 24-hour, Intragastric pH Following Daily Oral Dose Administration of RAB ER 50-mg Capsules Compared With Esomeprazole (Nexium) 40-mg Capsules and Rabeprazole (Aciphex) 20-mg Tablets to H. Pylori-Negative Healthy Subjects in a 5-day Treatment Regimen
Brief Title: A Study to Evaluate the Effect on 24-hour, Intragastric pH of RAB ER 50-mg Capsules Compared With Esomeprazole (Nexium) 40 mg Capsules and Rabeprazole (Aciphex) 20-mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E3810-A001-038
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: rabeprazole; esomeprazole; h. pylori-negative; nocturnal acid breakthrough; intragastric pH, PK/PD; effect on gastric pH in healthy, H. pylori-Negative subjects
MeSH Terms: interventions — Rabeprazole; Esomeprazole

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: E3810
- 2 (Active Comparator)
  Interventions: Drug: Aciphex (rabeprazole)
- 3 (Active Comparator)
  Interventions: Drug: Nexium (esomeprazole)

INTERVENTIONS:
Drug: E3810 — RAB ER 50 mg capsule once per day on Days 1-5
  Arms: 1
Drug: Aciphex (rabeprazole) — Aciphex (rabeprazole) 20 mg tablet once per day on Days 1-5
  Arms: 2
Drug: Nexium (esomeprazole) — Nexium (esomeprazole) 40 mg capsule once per day on Days 1-5
  Arms: 3

SUMMARY:
This will be a randomized, open-label, single-center, 3-way crossover study in healthy subjects who are confirmed to be Helicobacter pylori (H. pylori)-negative. The study will consist of 3 study periods separated by a washout period of at least 7 days. Subjects will receive study drugs once daily for 5 days. Barring any safety concerns, subjects will be discharged from the study on Day 6 of Period 3 after completion of discharge procedures.

ELIGIBILITY:
Key inclusion:

* Healthy male and female subjects, including women of child-bearing potential, aged 18 to 55 years, inclusive
* Subjects who are able to tolerate the insertion and placement of a pH probe on 2 occasions per study period (Day -1 and Day 5)

Key Exclusion:

* Subjects who are H. pylori-positive
* Subjects who have a history of any gastrointestinal disorder or surgery likely to influence drug absorption (e.g., history of gastric resection)
* Known hypersensitivity to rabeprazole, esomeprazole, or related compounds or any ingredient in the formulations
* Other standard clinical pharmacology exclusion criteria for healthy volunteers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Percentage of time that intragastric pH remains >4 | 24-hr period post-dose on Day 5

SECONDARY OUTCOMES:
Percentage of day- and night-time periods with intragastric pH >4 | Days 1 and 5
Number and duration of nocturnal acid breakthrough (NAB) episodes | Days 1 and 5
Proportion of subjects with nocturnal acid breakthrough (NAB) episodes | Days 1 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Philip Miner, Principal Investigator — Oklahoma Foundation for Digestive Research, 1000 N. Lincoln, Suite 210, Oklahoma City, OK 73104 USA
Locations (1):
- Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma, United States